CLINICAL TRIAL: NCT02123225
Title: Is the STOP-BANG Predictive of Worsening Obstructive Sleep Apnea in the Early Postoperative Period in Patients Undergoing Total Joint Arthroplasty?
Brief Title: Is the STOP-BANG Predictive of Worsening OSA in the Early Postop Period in Patients Undergoing TJA?
Status: Completed | Type: Observational
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dennis Spence, Regional Director, Nursing Research, NAVMEDWEST Region, United States Naval Medical Center, San Diego
Other Study IDs: NMCSD.2013.0045
Record Dates: First submitted 2014-04-21; First posted 2014-04-25 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Obstructive Sleep Apnea; Total Knee Arthroplasty
Keywords: STOP-BANG; Obstructive sleep apnea (OSA); total knee arthroplasty (TKA); portable monitoring; sleep medicine; unattended sleep study; postoperative sleep study
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to determine if the investigators can use the STOP-BANG score to identify those patients at risk for worsening Obstructive Sleep Apnea (OSA) symptoms in the early postoperative period after major surgery.

Hypotheses:

1. - Postoperative sleep apnea parameters will be worse when compared to baseline in patients with higher scores on the STOP-BANG.
2. - A higher STOP-BANG score will be predictive of worsening sleep apnea parameters in patients undergoing Total Knee Arthroscopy (TKA).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is associated with increased morbidity and mortality after total knee arthroplasty (TKA). Up to 30% of surgical patients have undiagnosed OSA; however, many patients are unable to obtain a sleep study prior to surgery. In recent years the STOP-BANG questionnaire (8 yes-no questions; ≥3 high-risk OSA) has become one of the most common tools used in the preoperative period to identify patients at high-risk for OSA. However, further research is needed to determine if the STOP-BANG is predictive of worsening of sleep apnea parameters in patients undergoing TKA.

The purpose of this prospective observational cohort study is to determine in TKA patients if the score on the STOP-BANG (<3, ≥3 to <5, or ≥5) is predictive of worsening sleep apnea parameters (AHI, time with SPO2 <90% & 85% [T90 & T85], lowest oxygen saturation [LSAT], & number of central apneas) during the first three days after surgery. The investigators propose to enroll N = 168 patients undergoing TKA at NMCSD who are receiving multimodal anesthesia/analgesia for surgery. Patients will complete a baseline unattended sleep study prior to surgery then again for the first three days after surgery. Patients will be categorized into three groups based on their STOP-BANG score (<3, ≥3 to <5, or ≥5) and the investigators will first compare the groups to identify if there are differences between baseline and postoperative sleep apnea parameters based on the STOP-BANG groups (<3, ≥3 to <5, or ≥5). If differences are found the investigators will use multiple regression analysis to determine if the STOP-BANG scores or categories and/or other covariates (i.e., comorbidity index, total morphine equivalents) are predictive of worsening sleep apnea during the first three days after surgery.

Results of this study may help improve patient safety by allowing us to identify which group of TKA patients with undiagnosed OSA may require more intensive postoperative monitoring and therapy (i.e, ICU admission, need for continuous end-tidal CO2 monitoring, postoperative positive airway pressure therapy) or change in the analgesic plan.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Scheduled for primary or revision TKA
* Able to read and understand the consent
* Able to complete an unattended OSA PM examination at home 1-60 days prior to surgery and for three days postoperatively

Exclusion Criteria:

* Polysomnography confirmed OSA
* Significant comorbid medical conditions that may degrade the accuracy of PM (moderate to severe pulmonary disease, neuromuscular disease, or congestive heart failure)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population will be N = 168 patients scheduled for primary or revision TKA between the ages of 18-90, at Naval Medical Center San Diego.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2013-12; Primary Completion 2016-11 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index | Baseline through postoperative night 3
  Measuring changes in the apnea hypopnea index on postoperative nights 1, 2, and 3 with unattended polysomnography.

SECONDARY OUTCOMES:
Change in time with oxygen saturation <85% | Baseline through postoperative night 3
  Measuring changes in the total time with oxygen saturations <85% on postoperative nights 1, 2 & 3 with unattended polysomnography.
Change in time with oxygen saturation <90% | Baseline through postoperative night 3
  Measuring changes in the total time with oxygen saturations <90% on postoperative nights 1, 2 & 3 with unattended polysomnography.

OTHER OUTCOMES:
Change in number of central apneas | Baseline through postoperative night 3
  Measuring changes in the total time number of central apnea episodes with unattended polysomnography between postoperative nights, 1,2, and 3.
Composite Complication Rate | 6 weeks postoperatively
  Defined as the incidence of composite complications: myocardial ishchemia or infarction, EKG changes, pulmonary embolism, need for CPAP, unplanned intubation, ICU admission, difficult intubation, pneumonia, or ARDS. Medical records will be reviewed to determine incidence of these complications through 6 weeks postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Spence, PhD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No